CLINICAL TRIAL: NCT01064648
Title: A Phase I/Randomized Phase II Study of Cediranib (NSC#732208) Versus Placebo in Combination With Cisplatin and Pemetrexed in Chemonaive Patients With Malignant Pleural Mesothelioma
Brief Title: Pemetrexed Disodium and Cisplatin With or Without Cediranib Maleate in Treating Patients With Malignant Pleural Mesothelioma
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NCI-2011-02015; NCI-2011-02015 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000665415; S0905; S0905 (Other: SWOG); S0905 (Other: CTEP); U10CA032102 (NIH); U10CA180830 (NIH); U10CA180888 (NIH)
Record Dates: First submitted 2010-02-05; First posted 2010-02-08 (Estimated); Results first posted 2020-02-05 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Epithelioid Mesothelioma; Pleural Malignant Mesothelioma; Recurrent Malignant Mesothelioma; Sarcomatoid Mesothelioma
MeSH Terms: conditions — Mesothelioma, Malignant; Solitary Fibrous Tumor, Pleural | interventions — cediranib; Cisplatin; 1,2-diaminocyclohexaneplatinum II citrate; Platinum; Pemetrexed

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm I (pemetrexed disodium, cisplatin, cediranib maleate)) (Experimental): Patients receive pemetrexed disodium IV over 10 minutes and cisplatin IV over 2 hours on day 1 and cediranib maleate PO QD on days 1-21. Treatment repeats every 21 days for 6 courses in the absence of disease progression or unacceptable toxicity. Patients then receive cediranib maleate alone PO QD in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Cediranib Maleate; Drug: Cisplatin; Other: Laboratory Biomarker Analysis; Drug: Pemetrexed Disodium
- Arm II (pemetrexed disodium, cisplatin, placebo) (Active Comparator): Patients receive pemetrexed disodium and cisplatin as in arm I and placebo PO QD on days 1-21. Treatment repeats every 21 days for 6 courses in the absence of disease progression or unacceptable toxicity. Patients then receive placebo alone PO QD in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Cisplatin; Other: Laboratory Biomarker Analysis; Drug: Pemetrexed Disodium; Other: Placebo Administration

INTERVENTIONS:
Drug: Cediranib Maleate — Given orally
  Other Names: AZD2171; AZD2171 Maleate; Recentin
  Arms: Arm I (pemetrexed disodium, cisplatin, cediranib maleate))
Drug: Cisplatin — Given IV
  Other Names: Abiplatin; Blastolem; Briplatin; CDDP; Cis-diammine-dichloroplatinum; Cis-diamminedichloridoplatinum; Cis-diamminedichloro Platinum (II); Cis-diamminedichloroplatinum; Cis-dichloroammine Platinum (II); Cis-platinous Diamine Dichloride; Cis-platinum; Cis-platinum II; Cis-platinum II Diamine Dichloride; Cismaplat; Cisplatina; Cisplatinum; Cisplatyl; Citoplatino; Citosin; Cysplatyna; DDP; Lederplatin; Metaplatin; Neoplatin; Peyrone's Chloride; Peyrone's Salt; Placis; Plastistil; Platamine; Platiblastin; Platiblastin-S; Platinex; Platinol; Platinol- AQ; Platinol-AQ; Platinol-AQ VHA Plus; Platinoxan; Platinum; Platinum Diamminodichloride; Platiran; Platistin; Platosin
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Pemetrexed Disodium — Given IV
  Other Names: Alimta; Almita; LY231514; N-[4-[2-(2-Amino-4,7-dihydro-4-oxo-1H-pyrrolo[2,3-d]pyrimidin-5-yl)ethyl]benzoyl]-L-glutamic Acid Disodium Salt
Other: Placebo Administration — Given orally
  Arms: Arm II (pemetrexed disodium, cisplatin, placebo)

SUMMARY:
This randomized phase I/II trial is studying the side effects and best dose of cediranib maleate when given together with pemetrexed disodium and cisplatin and to see how well it works in treating patients with malignant pleural mesothelioma. Drugs used in chemotherapy, pemetrexed disodium and cisplatin, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Cediranib maleate may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth and by blocking blood flow to the tumor. Giving pemetrexed disodium and cisplatin together with cediranib maleate may kill more tumor cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To establish the maximum tolerated dose (MTD) and the recommended phase II dose of cediranib maleate (cediranib) in combination with cisplatin and pemetrexed disodium (pemetrexed). (Phase I) II. To assess the safety and toxicity of the regimen. (Phase I) III. To assess whether cisplatin/pemetrexed plus cediranib as compared to cisplatin/pemetrexed plus placebo improves progression-free survival in patients with malignant pleural mesothelioma. (Phase II) IV. To compare overall survival in patients treated with cisplatin/pemetrexed plus cediranib to those treated with cisplatin/pemetrexed plus placebo. (Phase II) V. To assess the safety and toxicity profile of the regimen. (Phase II) VI. To assess response rate (confirmed and unconfirmed, complete and partial responses) and disease control rate (response or stable disease) in the subset of patients with measurable disease by Response Evaluation Criteria in Solid Tumors (RECIST) criteria. (Phase II) VII. To assess response rate and disease control rate using modified RECIST criteria for pleural tumors in the subset of patients with measurable disease by modified RECIST criteria for pleural tumors. (Phase II) VIII. To assess the rate of agreement between local and central pathology review of mesothelioma and its histologic subtypes. (Phase II) IX. To collect specimens for banking for use in future research studies. (Phase II)

OUTLINE: This is a phase I dose-escalation study of cediranib maleate followed by a phase II study.

PHASE I (CLOSED): Patients receive pemetrexed disodium intravenously (IV) over 10 minutes and cisplatin IV over 2 hours on day 1 and cediranib maleate orally (PO) once daily (QD) on days 1-21. Treatment repeats every 21 days for 6 courses in the absence of disease progression or unacceptable toxicity. Patients then receive cediranib maleate alone PO QD in the absence of disease progression or unacceptable toxicity.

PHASE II: Patients are randomized to 1 of 2 treatment arms.

ARM I: Patients receive pemetrexed disodium IV over 10 minutes and cisplatin IV over 2 hours on day 1 and cediranib maleate PO QD on days 1-21. Treatment repeats every 21 days for 6 courses in the absence of disease progression or unacceptable toxicity. Patients then receive cediranib maleate alone PO QD in the absence of disease progression or unacceptable toxicity.

ARM II: Patients receive pemetrexed disodium and cisplatin as in arm I and placebo PO QD on days 1-21. Treatment repeats every 21 days for 6 courses in the absence of disease progression or unacceptable toxicity. Patients then receive placebo alone PO QD in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 6 months for 2 years and then at 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Patient must have histologically or cytologically confirmed diagnosis of malignant pleural mesothelioma; surgical resection must not be planned
* Patients must have measurable or non-measurable disease by both RECIST and modified RECIST criteria for pleural tumors as documented by computed tomography (CT) scan; examinations for assessment of measurable disease must have been completed within 28 days prior to registration; examinations for assessment of non-measurable disease must have been performed within 42 days prior to registration; all disease must be assessed and documented on the RECIST 1.1 and Modified RECIST Baseline Tumor Assessment Form
* Patients must not have received any prior systemic therapy (chemotherapy or other biologic therapy) for their unresectable malignant pleural mesothelioma; prior systemic chemotherapy or biologic therapy is allowed as neoadjuvant or adjuvant treatment, disease has now recurred, and all systemic treatment was completed > 6 months prior registration; prior therapy must not have included cediranib
* Patients may have received prior surgery (e.g., pleurectomy, pleurodeisis) provided at least 28 days have elapsed since surgery (thoracic or other major surgeries) and patients have recovered from all associated toxicities at the time of registration; there must be no anticipated need for major surgical procedures during protocol treatment
* Patients may have received prior radiation therapy provided at least 28 days have elapsed since the last treatment and patients have recovered from all associated toxicities at the time of registration
* Institutions must seek additional patient consent for the banking and future use of specimens
* Patient must have Zubrod performance status 0-2
* Absolute neutrophil count >= 1,500 mcl
* Platelets >= 100,000/ml
* Hemoglobin >= 9.0 g/dl (may be reached by transfusion)
* Total bilirubin =< 1.5 x institutional upper limit of normal (IULN)
* Serum glutamic oxaloacetic transaminase (SGOT) or serum glutamate pyruvate transaminase (SGPT) =< 2.5 x ULN (if liver metastases are present, SGOT or SGPT must be =< 5.0 x IULN)
* Serum creatinine =< 1.5 x IULN
* Calculated creatinine clearance >= 60 mL/min
* Urine protein must be screened by urine analysis within 28 days prior to registration; patient must not have greater than +1 proteinuria on two consecutive dipsticks taken no less than 7 days apart; however, if the first urinalysis shows no protein, then a repeat urinalysis is not required
* Patient must have an electrocardiogram (ECG) performed within 42 days prior to registration; patient must not have mean corrected QT (QTc) > 500 msec (with Bazett's correction) in screening electrocardiogram, or other significant ECG abnormality, New York Heart Association (NYHA) classification III or IV; patient must not require concurrent use of drugs or biologics with proarrhythmic potential
* Patient must not be receiving any medication that may markedly affect renal function (e.g., vancomycin, amphotericin, pentamidine)
* Patient must not have had clinically significant hemoptysis, defined as greater than 1 tablespoon of bright red blood, within one year prior to registration; although hemoptysis has not been associated with cediranib, it may be a class effect for anti-angiogenic agents and therefore a risk factor for this experimental agent
* Patient must be able to swallow oral medications
* Patients must not have known human immunodeficiency virus (HIV) infection
* Patients must not be pregnant or nursing; women/men of reproductive potential must have agreed to use an effective contraceptive method; a woman is considered to be of "reproductive potential" if she has had menses at any time in the preceding 12 consecutive months; in addition to routine contraceptive methods, "effective contraception" also includes heterosexual celibacy and surgery intended to prevent pregnancy (or with a side-effect of pregnancy prevention) defined as a hysterectomy, bilateral oophorectomy or bilateral tubal ligation; however, if at any point a previously celibate patient chooses to become heterosexually active during the time period for use of contraceptive measures outlined in the protocol, he/she is responsible for beginning contraceptive measures
* Patient must have no plans to receive concurrent chemotherapy, hormonal therapy, radiotherapy, immunotherapy or any other type of therapy for treatment of cancer while on this protocol treatment
* No other prior malignancy is allowed except for the following: adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, adequately treated stage I or II cancer from which the patient is currently in complete remission, or any other cancer from which the patient has been disease free for five years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 117 (Actual)
Dates: Start 2010-03-15 (Actual); Primary Completion 2018-06-01 (Actual); Study Completion 2026-03-19 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Anne S Tsao, Principal Investigator — SWOG Cancer Research Network
Locations (231):
- United States (231):
  - Highlands Oncology Group - Rogers, Rogers, Arkansas
  - Kaiser Permanente-Deer Valley Medical Center, Antioch, California
  - Providence Saint Joseph Medical Center/Disney Family Cancer Center, Burbank, California
  - Kaiser Permanente-Fremont, Fremont, California
  - Kaiser Permanente-Fresno, Fresno, California
  - Los Angeles General Medical Center, Los Angeles, California
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California
  - Kaiser Permanente-Modesto, Modesto, California
  - Kaiser Permanente-Oakland, Oakland, California
  - UC Irvine Health/Chao Family Comprehensive Cancer Center, Orange, California
  - Kaiser Permanente-Redwood City, Redwood City, California
  - Kaiser Permanente-Richmond, Richmond, California
  - Kaiser Permanente-Roseville, Roseville, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - Kaiser Permanente-South Sacramento, Sacramento, California
  - Kaiser Permanente Sacramento Medical Center, Sacramento, California
  - Kaiser Permanente-San Francisco, San Francisco, California
  - Kaiser Permanente-Santa Teresa-San Jose, San Jose, California
  - Kaiser Permanente San Leandro, San Leandro, California
  - Kaiser Permanente-San Rafael, San Rafael, California
  - Kaiser Permanente Medical Center - Santa Clara, Santa Clara, California
  - Kaiser Permanente-Santa Rosa, Santa Rosa, California
  - Kaiser Permanente-South San Francisco, South San Francisco, California
  - Kaiser Permanente-Stockton, Stockton, California
  - Kaiser Permanente Medical Center-Vacaville, Vacaville, California
  - Kaiser Permanente-Vallejo, Vallejo, California
  - Kaiser Permanente-Walnut Creek, Walnut Creek, California
  - Smilow Cancer Hospital Care Center at Saint Francis, Hartford, Connecticut
  - Orlando Health Cancer Institute, Orlando, Florida
  - Northeast Georgia Medical Center-Gainesville, Gainesville, Georgia
  - Hawaii Cancer Care Inc - Waterfront Plaza, Honolulu, Hawaii
  - Queen's Medical Center, Honolulu, Hawaii
  - Straub Clinic and Hospital, Honolulu, Hawaii
  - University of Hawaii Cancer Center, Honolulu, Hawaii
  - Hawaii Cancer Care Inc-Liliha, Honolulu, Hawaii
  - Kuakini Medical Center, Honolulu, Hawaii
  - Queen's Cancer Center - Kuakini, Honolulu, Hawaii
  - Kaiser Permanente Moanalua Medical Center, Honolulu, Hawaii
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Castle Medical Center, Kailua, Hawaii
  - Wilcox Memorial Hospital and Kauai Medical Clinic, Lihue, Hawaii
  - Pali Momi Medical Center, ‘Aiea, Hawaii
  - Queen's Cancer Center - Pearlridge, ‘Aiea, Hawaii
  - Saint Alphonsus Cancer Care Center-Boise, Boise, Idaho
  - Kootenai Health - Coeur d'Alene, Coeur d'Alene, Idaho
  - Kootenai Clinic Cancer Services - Post Falls, Post Falls, Idaho
  - Kootenai Clinic Cancer Services - Sandpoint, Sandpoint, Idaho
  - OSF Saint Joseph Medical Center, Bloomington, Illinois
  - Illinois CancerCare-Bloomington, Bloomington, Illinois
  - Illinois CancerCare-Canton, Canton, Illinois
  - Memorial Hospital of Carbondale, Carbondale, Illinois
  - Illinois CancerCare-Carthage, Carthage, Illinois
  - Centralia Oncology Clinic, Centralia, Illinois
  - Cancer Care Specialists of Illinois - Decatur, Decatur, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Heartland Cancer Research NCORP, Decatur, Illinois
  - Crossroads Cancer Center, Effingham, Illinois
  - Illinois CancerCare-Eureka, Eureka, Illinois
  - Illinois CancerCare-Galesburg, Galesburg, Illinois
  - Western Illinois Cancer Treatment Center, Galesburg, Illinois
  - Illinois CancerCare-Kewanee Clinic, Kewanee, Illinois
  - Illinois CancerCare-Macomb, Macomb, Illinois
  - Cancer Care Center of O'Fallon, O'Fallon, Illinois
  - Illinois CancerCare-Ottawa Clinic, Ottawa, Illinois
  - Radiation Oncology of Northern Illinois, Ottawa, Illinois
  - Illinois CancerCare-Pekin, Pekin, Illinois
  - OSF Saint Francis Radiation Oncology at Pekin, Pekin, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - OSF Saint Francis Radiation Oncology at Peoria Cancer Center, Peoria, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - OSF Saint Francis Medical Center, Peoria, Illinois
  - Illinois CancerCare-Peru, Peru, Illinois
  - Valley Radiation Oncology, Peru, Illinois
  - Illinois CancerCare-Princeton, Princeton, Illinois
  - Central Illinois Hematology Oncology Center, Springfield, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Springfield Clinic, Springfield, Illinois
  - Springfield Memorial Hospital, Springfield, Illinois
  - Franciscan Saint Francis Health-Beech Grove, Beech Grove, Indiana
  - Franciscan Health Indianapolis, Indianapolis, Indiana
  - Reid Health, Richmond, Indiana
  - Cotton O'Neil Cancer Center / Stormont Vail Health, Topeka, Kansas
  - Oncology Hematology Care Inc-Crestview, Crestview Hills, Kentucky
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - Michigan Cancer Research Consortium NCORP, Ann Arbor, Michigan
  - Trinity Health Saint Joseph Mercy Hospital Ann Arbor, Ann Arbor, Michigan
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Corewell Health Dearborn Hospital, Dearborn, Michigan
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - Henry Ford Health Saint John Hospital, Detroit, Michigan
  - Weisberg Cancer Treatment Center, Farmington Hills, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Genesys Regional Medical Center-West Flint Campus, Flint, Michigan
  - Allegiance Health, Jackson, Michigan
  - University of Michigan Health - Sparrow Lansing, Lansing, Michigan
  - Trinity Health Saint Mary Mercy Livonia Hospital, Livonia, Michigan
  - Trinity Health Saint Joseph Mercy Oakland Hospital, Pontiac, Michigan
  - Lake Huron Medical Center, Port Huron, Michigan
  - MyMichigan Medical Center Saginaw, Saginaw, Michigan
  - Henry Ford Health Warren Hospital, Warren, Michigan
  - Singing River Hospital, Pascagoula, Mississippi
  - Parkland Health Center-Bonne Terre, Bonne Terre, Missouri
  - Mercy Cancer Center - Cape Girardeau, Cape Girardeau, Missouri
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - MU Health Care Goldschmidt Cancer Center, Jefferson City, Missouri
  - Sainte Genevieve County Memorial Hospital, Sainte Genevieve, Missouri
  - Missouri Baptist Medical Center, St Louis, Missouri
  - Missouri Baptist Sullivan Hospital, Sullivan, Missouri
  - BJC Outpatient Center at Sunset Hills, Sunset Hills, Missouri
  - Community Hospital of Anaconda, Anaconda, Montana
  - Billings Clinic Cancer Center, Billings, Montana
  - Saint Vincent Healthcare, Billings, Montana
  - Montana Cancer Consortium NCORP, Billings, Montana
  - Saint Vincent Frontier Cancer Center, Billings, Montana
  - Bozeman Health Deaconess Hospital, Bozeman, Montana
  - Saint James Community Hospital and Cancer Treatment Center, Butte, Montana
  - Benefis Sletten Cancer Institute, Great Falls, Montana
  - Great Falls Clinic, Great Falls, Montana
  - Saint Peter's Community Hospital, Helena, Montana
  - Glacier Oncology PLLC, Kalispell, Montana
  - Logan Health Medical Center, Kalispell, Montana
  - Montana Cancer Specialists, Missoula, Montana
  - Saint Patrick Hospital - Community Hospital, Missoula, Montana
  - Community Medical Center, Missoula, Montana
  - Novant Health Presbyterian Medical Center, Charlotte, North Carolina
  - Novant Health Carolina Surgical - Randolph, Charlotte, North Carolina
  - Oncology Specialists of Charlotte, Charlotte, North Carolina
  - Southern Oncology Specialists-Charlotte, Charlotte, North Carolina
  - Margaret R Pardee Memorial Hospital, Hendersonville, North Carolina
  - Novant Health Cancer Institute - Huntersville, Huntersville, North Carolina
  - Southern Oncology Specialists-Huntersville, Huntersville, North Carolina
  - Matthews Radiation Oncology Center, Matthews, North Carolina
  - Novant Health Cancer Institute - Matthews, Matthews, North Carolina
  - Novant Health Cancer Institute - Mooresville, Mooresville, North Carolina
  - Iredell Memorial Hospital, Statesville, North Carolina
  - Southeast Clinical Oncology Research Consortium NCORP, Winston-Salem, North Carolina
  - Strecker Cancer Center-Belpre, Belpre, Ohio
  - Adena Regional Medical Center, Chillicothe, Ohio
  - Oncology Hematology Care Inc-Eden Park, Cincinnati, Ohio
  - Oncology Hematology Care Inc-Mercy West, Cincinnati, Ohio
  - Oncology Hematology Care Inc-Anderson, Cincinnati, Ohio
  - Oncology Hematology Care Inc-Kenwood, Cincinnati, Ohio
  - Oncology Hematology Care Inc-Blue Ash, Cincinnati, Ohio
  - Mount Carmel East Hospital, Columbus, Ohio
  - Columbus Oncology and Hematology Associates Inc, Columbus, Ohio
  - Riverside Methodist Hospital, Columbus, Ohio
  - Columbus NCI Community Oncology Research Program, Columbus, Ohio
  - Grant Medical Center, Columbus, Ohio
  - The Mark H Zangmeister Center, Columbus, Ohio
  - Mount Carmel Health Center West, Columbus, Ohio
  - Doctors Hospital, Columbus, Ohio
  - Grandview Hospital, Dayton, Ohio
  - Good Samaritan Hospital - Dayton, Dayton, Ohio
  - Miami Valley Hospital, Dayton, Ohio
  - Miami Valley Hospital North, Dayton, Ohio
  - Dayton NCI Community Oncology Research Program, Dayton, Ohio
  - Delaware Health Center-Grady Cancer Center, Delaware, Ohio
  - Delaware Radiation Oncology, Delaware, Ohio
  - Grady Memorial Hospital, Delaware, Ohio
  - Oncology Hematology Care Inc-Healthplex, Fairfield, Ohio
  - Blanchard Valley Hospital, Findlay, Ohio
  - Atrium Medical Center-Middletown Regional Hospital, Franklin, Ohio
  - Wayne Hospital, Greenville, Ohio
  - Kettering Medical Center, Kettering, Ohio
  - Fairfield Medical Center, Lancaster, Ohio
  - OhioHealth Mansfield Hospital, Mansfield, Ohio
  - Marietta Memorial Hospital, Marietta, Ohio
  - OhioHealth Marion General Hospital, Marion, Ohio
  - Knox Community Hospital, Mount Vernon, Ohio
  - Licking Memorial Hospital, Newark, Ohio
  - Newark Radiation Oncology, Newark, Ohio
  - Southern Ohio Medical Center, Portsmouth, Ohio
  - Springfield Regional Medical Center, Springfield, Ohio
  - Upper Valley Medical Center, Troy, Ohio
  - Saint Ann's Hospital, Westerville, Ohio
  - Greene Memorial Hospital, Xenia, Ohio
  - Genesis Healthcare System Cancer Care Center, Zanesville, Ohio
  - Clackamas Radiation Oncology Center, Clackamas, Oregon
  - Providence Milwaukie Hospital, Milwaukie, Oregon
  - Providence Newberg Medical Center, Newberg, Oregon
  - Providence Willamette Falls Medical Center, Oregon City, Oregon
  - Providence Portland Medical Center, Portland, Oregon
  - Providence Saint Vincent Medical Center, Portland, Oregon
  - Prisma Health Cancer Institute - Spartanburg, Boiling Springs, South Carolina
  - Prisma Health Cancer Institute - Easley, Easley, South Carolina
  - Greenville Health System Cancer Institute-Andrews, Greenville, South Carolina
  - Prisma Health Cancer Institute - Butternut, Greenville, South Carolina
  - Prisma Health Cancer Institute - Faris, Greenville, South Carolina
  - Prisma Health Greenville Memorial Hospital, Greenville, South Carolina
  - Prisma Health Cancer Institute - Eastside, Greenville, South Carolina
  - Prisma Health Cancer Institute - Greer, Greer, South Carolina
  - Prisma Health Cancer Institute - Seneca, Seneca, South Carolina
  - Bristol Regional Medical Center, Bristol, Tennessee
  - Wellmont Medical Associates Oncology and Hematology-Bristol, Bristol, Tennessee
  - Wellmont Medical Associates Oncology and Hematology-Johnson City, Johnson City, Tennessee
  - Ballad Health Cancer Care - Kingsport, Kingsport, Tennessee
  - Wellmont Holston Valley Hospital and Medical Center, Kingsport, Tennessee
  - M D Anderson Cancer Center, Houston, Texas
  - Danville Regional Medical Center, Danville, Virginia
  - Ballad Health Cancer Care - Norton, Norton, Virginia
  - Cancer Care Center at Island Hospital, Anacortes, Washington
  - PeaceHealth Saint Joseph Medical Center, Bellingham, Washington
  - Highline Medical Center-Main Campus, Burien, Washington
  - Swedish Cancer Institute-Edmonds, Edmonds, Washington
  - Swedish Cancer Institute-Issaquah, Issaquah, Washington
  - Kadlec Clinic Hematology and Oncology, Kennewick, Washington
  - FHCC at EvergreenHealth, Kirkland, Washington
  - PeaceHealth Saint John Medical Center, Longview, Washington
  - Skagit Valley Hospital, Mount Vernon, Washington
  - Harrison HealthPartners Hematology and Oncology-Poulsbo, Poulsbo, Washington
  - Harborview Medical Center, Seattle, Washington
  - Minor and James Medical PLLC, Seattle, Washington
  - Swedish Medical Center-Ballard Campus, Seattle, Washington
  - Fred Hutchinson Cancer Center, Seattle, Washington
  - Kaiser Permanente Washington, Seattle, Washington
  - Swedish Medical Center-First Hill, Seattle, Washington
  - University of Washington Medical Center - Montlake, Seattle, Washington
  - PeaceHealth United General Medical Center, Sedro-Woolley, Washington
  - Saint Michael Cancer Center, Silverdale, Washington
  - Cancer Care Northwest - Spokane South, Spokane, Washington
  - Evergreen Hematology and Oncology PS, Spokane, Washington
  - Rockwood Clinic, Spokane, Washington
  - PeaceHealth Southwest Medical Center, Vancouver, Washington
  - Compass Oncology Vancouver, Vancouver, Washington
  - Wenatchee Valley Hospital and Clinics, Wenatchee, Washington
  - Rocky Mountain Oncology, Casper, Wyoming
  - Big Horn Basin Cancer Center, Cody, Wyoming
  - Billings Clinic-Cody, Cody, Wyoming
  - Welch Cancer Center, Sheridan, Wyoming

REFERENCES:
- [Derived] Tsao AS, Miao J, Wistuba II, Vogelzang NJ, Heymach JV, Fossella FV, Lu C, Velasco MR, Box-Noriega B, Hueftle JG, Gadgeel S, Redman MW, Gandara DR, Kelly K. Phase II Trial of Cediranib in Combination With Cisplatin and Pemetrexed in Chemotherapy-Naive Patients With Unresectable Malignant Pleural Mesothelioma (SWOG S0905). J Clin Oncol. 2019 Oct 1;37(28):2537-2547. doi: 10.1200/JCO.19.00269. Epub 2019 Aug 6. PMID 31386610

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 117 participants were enrolled, only 112 participants were included in the analysis: 5 patients were either not eligible or not analyzable. Thus these 5 patients were excluded from any analysis.
Groups:
- Phase I Cisplatin-pemetrexed Cediranib 30mg; Phase II Cisplatin-pemetrexed Cediranib 20mg: Patients receive pemetrexed disodium IV over 10 minutes and cisplatin IV over 2 hours on day 1 and cediranib maleate PO QD on days 1-21. Treatment repeats every 21 days for 6 courses in the absence of disease progression or unacceptable toxicity. Patients then receive cediranib maleate alone PO QD in the absence of disease progression or unacceptable toxicity.
  Cediranib Maleate: Given orally
  Cisplatin: Given IV
  Laboratory Biomarker Analysis: Correlative studies
  Pemetrexed Disodium: Given IV
- Phase I Cisplatin-pemetrexed Cediranib 20mg: Patients receive pemetrexed disodium and cisplatin as in arm I and placebo PO QD on days 1-21. Treatment repeats every 21 days for 6 courses in the absence of disease progression or unacceptable toxicity. Patients then receive placebo alone PO QD in the absence of disease progression or unacceptable toxicity.
  Cisplatin: Given IV
  Laboratory Biomarker Analysis: Correlative studies
  Pemetrexed Disodium: Given IV
  Placebo: Given orally
- Phase II Cisplatin-pemetrexed Placebo: Patients receive pemetrexed disodium IV over 10 minutes and cisplatin IV over 2 hours on day 1 and placebo PO QD on days 1-21. Treatment repeats every 21 days for 6 courses in the absence of disease progression or unacceptable toxicity. Patients then receive placebo alone PO QD in the absence of disease progression or unacceptable toxicity.
  Placebo: Given orally
  Cisplatin: Given IV
  Laboratory Biomarker Analysis: Correlative studies
  Pemetrexed Disodium: Given IV
Period: Phase I Cohort1: Dose Level 1
Arm/Group | Phase I Cisplatin-pemetrexed Cediranib 30mg | Phase I Cisplatin-pemetrexed Cediranib 20mg | Phase II Cisplatin-pemetrexed Cediranib 20mg | Phase II Cisplatin-pemetrexed Placebo
Started | 7 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0
Not Completed | 7 | 0 | 0 | 0
Not completed — Progression | 5 | 0 | 0 | 0
Not completed — Non-protocol specified | 2 | 0 | 0 | 0
Period: Phase I Cohort 2: Dose Level 2
Arm/Group | Phase I Cisplatin-pemetrexed Cediranib 30mg | Phase I Cisplatin-pemetrexed Cediranib 20mg | Phase II Cisplatin-pemetrexed Cediranib 20mg | Phase II Cisplatin-pemetrexed Placebo
Started | 0 | 13 | 0 | 0
Completed | 0 | 0 | 0 | 0
Not Completed | 0 | 13 | 0 | 0
Not completed — Adverse Event | 0 | 3 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0
Not completed — Progression | 0 | 5 | 0 | 0
Not completed — Non-protocol specified | 0 | 4 | 0 | 0
Period: Phase II
Arm/Group | Phase I Cisplatin-pemetrexed Cediranib 30mg | Phase I Cisplatin-pemetrexed Cediranib 20mg | Phase II Cisplatin-pemetrexed Cediranib 20mg | Phase II Cisplatin-pemetrexed Placebo
Started | 0 | 0 | 49 | 48
Completed | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 49 | 48
Not completed — Adverse Event | 0 | 0 | 15 | 8
Not completed — Death | 0 | 0 | 4 | 5
Not completed — Withdrawal by Subject | 0 | 0 | 2 | 5
Not completed — Progression | 0 | 0 | 21 | 27
Not completed — Non-protocol specified | 0 | 0 | 5 | 3
Not completed — Under Review | 0 | 0 | 2 | 0

BASELINE CHARACTERISTICS:
Population: 117 participants were enrolled, only 112 participants were included in the analysis: 5 patients were either not eligible or not analyzable. Thus these 5 patients were excluded from any analysis.
Groups:
- Phase I All Participants: All participants from Phase I
- Total: Total of all reporting groups
Arm/Group | Phase I All Participants | Phase II Cisplatin-pemetrexed Cediranib 20mg | Phase II Cisplatin-pemetrexed Placebo | Total
Number analyzed (Participants) | 20 | 45 | 47 | 112
Age, Continuous [Median (Full Range); unit: years] | 64.4 [43.6 to 83.6] | 71.3 [45.5 to 82.1] | 71.8 [50.9 to 85.3] | 69.8 [43.6 to 85.3]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 7 | 7 | 19
  Male | 15 | 38 | 40 | 93
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 3 | 2 | 6
  Not Hispanic or Latino | 19 | 41 | 44 | 104
  Unknown or Not Reported | 0 | 1 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 2 | 0 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 2 | 1 | 3 | 6
  White | 15 | 43 | 42 | 100
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 2 | 4
Zubrod Performance Status [Count of Participants; unit: Participants] — Patients will be graded according to the Zubrod Performance Status Scale:
  0: Fully active, able to carry on all pre-disease performance without restriction.
  1. Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light housework, office work.
  2. Ambulatory and capable of self-care but unable to carry out any work activities; up and about more than 50% of waking hours.
  The higher grade is, the worse performance status is.
  Participants
    0-1 | 19 | 42 | 44 | 105
    2 | 1 | 3 | 3 | 7
Histology [Count of Participants; unit: Participants]
  Epitheliod or mesothelioma, NOS | 18 | 34 | 35 | 87
  Biphasic or sarcomatoid | 2 | 11 | 12 | 25
Prior history of radiation [Count of Participants; unit: Participants]
  Yes | 5 | 8 | 9 | 22
  No | 15 | 37 | 38 | 90
Prior history of definitive surgery [Count of Participants; unit: Participants]
  Yes | 3 | 12 | 6 | 21
  No | 17 | 33 | 41 | 91
Measurable Disease per RECIST 1.1 [Count of Participants; unit: Participants]
  Measurable | 17 | 35 | 40 | 92
  Non-measurable | 3 | 10 | 7 | 20
Measurable Disease per Modified RECIST for Pleural Tumors [Count of Participants; unit: Participants]
  Measurable | 19 | 36 | 30 | 85
  Non-measurable | 1 | 9 | 17 | 27

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose of Cediranib in Combination With Cisplatin and Pemetrexed (Phase I)
Description: MTD was determined by testing dose-de-escalation to 20mg PO daily on dose de-escalation cohort 1 to 2 with 3 to 6 patients each. MTD reflects the highest dose of drug that did not cause a Dose-Limiting Toxicity (DLT) in > 33% of participants. Toxicities will be graded according to the CTEP Active Version of the NCI Common Terminology Criteria for Adverse Events. Dose-limiting toxicities (DLT) apply only during Cycle 1 and must be drug-related (i.e. possibly, probably or definitely related to one of the 3 study drugs). The following events occurring in the first cycle of treatment are considered dose limiting.
  1. Febrile neutropenia
  2. Grade 4 neutrophil count decrease for more than 7 days' duration
  3. Grade 4 platelet count decrease
  4. Grade 3 or 4 non-hematologic toxicity (excluding alopecia)
Time Frame: Weekly during first cycle (1cycle = 21 days). Then will be reported every cycle while patient is on treatment.
Measure: Number; unit: mg
Groups:
- All Phase I Participants: All participants from Phase I who are eligible for DLT. Patients will be considered evaluable for DLT if they received at least 14 doses of cediranib at the assigned dose during Cycle 1 and at least one dose each of pemetrexed and cisplatin, or if they developed a DLT. If a patient does not develop a DLT but does not complete at least 14 doses of cediranib and one dose each of pemetrexed and cisplatin during Cycle 1 due to any reason, the patient will be considered not evaluable for DLT and will be replaced.
Arm/Group | All Phase I Participants
Number analyzed (Participants) | 20
mg | 20

2. Primary Outcome: Progression-free Survival (Phase II)
Description: From date of registration to date of first documentation of progression or symptomatic deterioration, or death due to any cause. Patients last known to be alive and progression free are censored at date of last contact. Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v 1.1), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesions, or the appearance of new lesions.
Time Frame: From date of registration to date of first documentation of progression or symptomatic deterioration, or death due to any cause, whichever came first, assessed up to 5 years.Disease assessment will be repeated every 6 weeks until disease progression.
Population: Only eligible and analyzable patients were included.
Measure: Median (95% Confidence Interval); unit: month
Arm/Group | Phase II Cisplatin-pemetrexed Cediranib 20mg | Phase II Cisplatin-pemetrexed Placebo
Number analyzed (Participants) | 45 | 47
month | 7.2 [5.5 to 8.5] | 5.6 [4.6 to 6.2]
Statistical Analysis 1: Comparison: Phase II Cisplatin-pemetrexed Cediranib 20mg vs Phase II Cisplatin-pemetrexed Placebo; Test type: Other; p = 0.06, Log Rank — 1-sided p-value; Stratified log rank test by performance status and histology type; Hazard Ratio (HR) = 0.71, 80% CI 2-sided [0.54 to 0.95]

3. Secondary Outcome: Overall Survival (Phase II)
Description: From date of registration to date of death due to any cause. Patients last known to be alive are censored at date of last contact.
Time Frame: From date of registration to death.Disease assessment will be repeated every 6 weeks until disease progression. After progression, follow up will occur every 6 months for the first two years and then at the end of the third year after registration.
Population: Only eligible and analyzable patients are included in the analysis.
Measure: Median (95% Confidence Interval); unit: month
Arm/Group | Phase II Cisplatin-pemetrexed Cediranib 20mg | Phase II Cisplatin-pemetrexed Placebo
Number analyzed (Participants) | 45 | 47
month | 10 [7.7 to 13.5] | 8.5 [6.6 to 13.8]
Statistical Analysis 1: Comparison: Phase II Cisplatin-pemetrexed Cediranib 20mg vs Phase II Cisplatin-pemetrexed Placebo; Test type: Other; p = 0.28, Log Rank — 1-sided p-value; Stratified log-rank test by performance status and histology; Hazard Ratio (HR) = 0.88, 80% CI 2-sided [0.65 to 1.17]

4. Secondary Outcome: Response Rate by RECIST1.1 (Phase II)
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1): Complete Response (CR), Disappearance of all measurable and non-measurable disease; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
  All target measurable lesions must be assessed using the same techniques as baseline.
Time Frame: Disease assessment will be repeated every 6 weeks until disease progression, up to 3 years. Best response is documented for as long as the patient remains on protocol treatment.
Population: Only eligible patients with baseline measurable disease per RECIST 1.1 were included in the analysis.
Measure: Number (95% Confidence Interval); unit: percentage of analyzed participants
Arm/Group | Phase II Cisplatin-pemetrexed Cediranib 20mg | Phase II Cisplatin-pemetrexed Placebo
Number analyzed (Participants) | 35 | 40
percentage of analyzed participants | 26 [12 to 43] | 15 [6 to 30]
Statistical Analysis 1: Comparison: Phase II Cisplatin-pemetrexed Cediranib 20mg vs Phase II Cisplatin-pemetrexed Placebo; Test type: Other; p = 0.15, Chi-squared — 1-sided p-value; Stratified Chi-square by performance status and histology; Odds Ratio (OR) = 1.85, 95% CI 2-sided [0.59 to 5.83]

5. Secondary Outcome: Disease Control Rate by RECIST 1.1 (Phase II)
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1): Complete Response (CR), Disappearance of all measurable and non-measurable disease; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Stable Disease (STA): Does not qualify for CR, PR, Progression or Symptomatic Deterioration. Disease Control Rate (DCR) = CR + PR + STA
  All target measurable lesions must be assessed using the same techniques as baseline.
Time Frame: Disease assessment will be repeated every 6 weeks until disease progression, up to 3 years.Disease control rate is documented for as long as the patient remains on protocol treatment.
Population: Eligible patients with baseline eligible disease per RECIST 1.1 were included in the analysis.
Measure: Number (95% Confidence Interval); unit: percentage of analyzed participants
Arm/Group | Phase II Cisplatin-pemetrexed Cediranib 20mg | Phase II Cisplatin-pemetrexed Placebo
Number analyzed (Participants) | 35 | 40
percentage of analyzed participants | 74 [57 to 88] | 80 [64 to 91]
Statistical Analysis 1: Comparison: Phase II Cisplatin-pemetrexed Cediranib 20mg vs Phase II Cisplatin-pemetrexed Placebo; Test type: Other; p = 0.09, Chi-squared — 1-sided p-value; Stratified Chi-Square by performance status and histology; Odds Ratio (OR) = 0.45, 95% CI 2-sided [0.14 to 1.49]

6. Secondary Outcome: Response Rate by Modified RECIST (Phase II)
Description: Per modified RECIST for Pleural Tumors. In addition to RECIST1.1, for modified RECIST, measurements based on the sum of 6 CT cuts in the pleural perpendicular to the chest wall are applied to standard RECIST criterial (sum of 6 = one univariate diameter). Complete Response (CR), Disappearance of all measurable and non-measurable disease; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
  All target measurable lesions must be assessed using the same techniques as baseline.
Time Frame: Disease assessment will be repeated every 6 weeks until disease progression, up to 3 years.Best response is documented for as long as the patient remains on protocol treatment.
Population: Eligible patients with baseline measurable disease per modified RECIST were included in the analysis.
Measure: Number (95% Confidence Interval); unit: percentage of analyzed participants
Arm/Group | Phase II Cisplatin-pemetrexed Cediranib 20mg | Phase II Cisplatin-pemetrexed Placebo
Number analyzed (Participants) | 36 | 30
percentage of analyzed participants | 50 [33 to 67] | 20 [8 to 39]
Statistical Analysis 1: Comparison: Phase II Cisplatin-pemetrexed Cediranib 20mg vs Phase II Cisplatin-pemetrexed Placebo; Test type: Other; p = 0.006, Chi-squared — 1-sided p-value; Stratified Chi-Square by performance status and histology; Odds Ratio (OR) = 4.3, 95% CI 2-sided [1.4 to 13.3]

7. Secondary Outcome: Disease Control Rate by Modified RECIST (Phase II)
Description: Per modified RECIST for Pleural Tumors. In addition to RECIST1.1, for modified RECIST, measurements based on the sum of 6 CT cuts in the pleural perpendicular to the chest wall are applied to standard RECIST criterial (sum of 6 = one univariate diameter). Complete Response (CR), Disappearance of all measurable and non-measurable disease; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Stable Disease (STA), does not qualify for CR, PR, Progression or Symptomatic Deterioration. Disease Control Rate (DCR) = CR + PR + STA.
  All target measurable lesions must be assessed using the same techniques as baseline.
Time Frame: Disease assessment will be repeated every 6 weeks until disease progression, up to 3 years.Disease control is documented for as long as the patient remains on protocol treatment.
Population: Eligible patients with baseline measurable disease per modified RECIST were included in the analysis.
Measure: Number (95% Confidence Interval); unit: percentage of analyzed participants
Arm/Group | Phase II Cisplatin-pemetrexed Cediranib 20mg | Phase II Cisplatin-pemetrexed Placebo
Number analyzed (Participants) | 36 | 30
percentage of analyzed participants | 75 [58 to 88] | 83 [65 to 94]
Statistical Analysis 1: Comparison: Phase II Cisplatin-pemetrexed Cediranib 20mg vs Phase II Cisplatin-pemetrexed Placebo; Test type: Other; p = 0.19, Chi-squared — 1-sided p-value; Stratified Chi-Square by performance status and histology; Odds Ratio (OR) = 0.59, 95% CI 2-sided [0.18 to 1.94]

8. Secondary Outcome: (Phase I) Number of Patients With Gr 3 Through 5 Adverse Events That Are Related to Study Drugs
Description: Adverse Events (AEs) are reported by CTCAE Version 4.0. Only adverse events that are possibly, probably or definitely related to study drug are reported.
Time Frame: Toxicity assessment is repeated weekly during first cycle (1cycle = 21 days), then every cycle while patient is on treatment.
Population: Patients who received at least one dose of protocol treatment.
Measure: Number; unit: Participants
Groups:
- Phase I Cisplatin-pemetrexed Cediranib 30mg: Phase I Cisplatin-pemetrexed Cediranib 30mg
- Phase I Cisplatin-pemetrexed Cediranib 20mg: Phase I Cisplatin-pemetrexed Cediranib 20mg
Arm/Group | Phase I Cisplatin-pemetrexed Cediranib 30mg | Phase I Cisplatin-pemetrexed Cediranib 20mg
Number analyzed (Participants) | 7 | 13
Participants
  Abdominal pain | 0 | 2
  Anemia | 0 | 1
  Constipation | 0 | 1
  Dehydration | 0 | 3
  Diarrhea | 2 | 2
  Dyspnea | 0 | 2
  Fatigue | 2 | 1
  Gastrointestinal disorders - Other, specify | 0 | 1
  Heart failure | 0 | 1
  Hypertension | 0 | 1
  Hypokalemia | 0 | 1
  Hypomagnesemia | 1 | 0
  Hyponatremia | 0 | 1
  Irregular menstruation | 0 | 1
  Lymphocyte count decreased | 2 | 0
  Mucositis oral | 0 | 1
  Nausea | 0 | 1
  Nervous system disorders - Other, specify | 0 | 1
  Neutrophil count decreased | 1 | 2
  Palmar-plantar erythrodysesthesia syndrome | 1 | 0
  Peripheral sensory neuropathy | 0 | 1
  Platelet count decreased | 0 | 3
  Pulmonary hypertension | 0 | 1
  Vomiting | 0 | 2
  Weight loss | 1 | 0
  White blood cell decreased | 0 | 1

9. Secondary Outcome: (Phase II) Number of Patients With Gr 3 Through 5 Adverse Events That Are Related to Study Drugs
Description: as for outcome 8
Time Frame: Toxicity assessment is repeated every 3 weeks while patient is on treatment.
Population: Patients who received at least one dose of protocol treatment.
Measure: Number; unit: Participants
Groups:
- Phase II Cisplatin-pemetrexed Cediranib 20mg: Phase II Cisplatin-pemetrexed Cediranib 20mg
- Phase II Cisplatin-pemetrexed Placebo: Phase II Cisplatin-pemetrexed Placebo
Arm/Group | Phase II Cisplatin-pemetrexed Cediranib 20mg | Phase II Cisplatin-pemetrexed Placebo
Number analyzed (Participants) | 44 | 44
Participants
  Acute coronary syndrome | 0 | 1
  Anemia | 1 | 7
  Anorexia | 7 | 4
  Atrial fibrillation | 2 | 0
  Atrial flutter | 1 | 1
  Chest wall pain | 0 | 1
  Creatinine increased | 0 | 1
  Death NOS | 1 | 0
  Dehydration | 4 | 2
  Delirium | 0 | 1
  Diarrhea | 2 | 0
  Duodenal hemorrhage | 0 | 1
  Dyspnea | 2 | 2
  Epistaxis | 1 | 0
  Fall | 1 | 0
  Fatigue | 6 | 5
  General disorders and admin site conditions-Other | 0 | 1
  Generalized muscle weakness | 1 | 1
  Glucose intolerance | 1 | 0
  Headache | 1 | 0
  Hearing impaired | 0 | 2
  Heart failure | 1 | 0
  Hyperglycemia | 1 | 0
  Hypertension | 9 | 0
  Hypocalcemia | 1 | 1
  Hypokalemia | 2 | 0
  Hypomagnesemia | 2 | 0
  Hyponatremia | 5 | 1
  Hypotension | 3 | 0
  Hypoxia | 0 | 1
  Intracranial hemorrhage | 1 | 0
  Lung infection | 1 | 1
  Lymphocyte count decreased | 2 | 2
  Mucositis oral | 1 | 0
  Nausea | 4 | 5
  Neutrophil count decreased | 6 | 8
  Non-cardiac chest pain | 1 | 0
  Peripheral sensory neuropathy | 0 | 1
  Platelet count decreased | 4 | 2
  Rash maculo-papular | 1 | 0
  Renal and urinary disorders - Other, specify | 0 | 1
  Respiratory failure | 2 | 0
  Seizure | 1 | 0
  Sinus bradycardia | 2 | 0
  Supraventricular tachycardia | 1 | 0
  Syncope | 0 | 1
  Thromboembolic event | 3 | 3
  Urinary tract infection | 0 | 1
  Vomiting | 0 | 2
  Weight loss | 4 | 0
  White blood cell decreased | 3 | 4
  Wound dehiscence | 1 | 0

ADVERSE EVENTS:
Time Frame: For phase I patients, adverse assessment is repeated weekly during first cycle (1 cycle = 21 days), then every cycle until patient is off protocol treatment. For phase II patients, adverse assessment is repeated every cycle until patient is off protocol treatment, up to 3 years.
Description: For Adverse Event assessment, we include patients who are eligible and evaluable for adverse events (e.g., received at least one dose of protocol treatment) in the analysis. For all-cause mortality, we include all eligible patients in the analysis.
Arm/Group | Phase I Cisplatin-pemetrexed Cediranib 30mg | Phase I Cisplatin-pemetrexed Cediranib 20mg | Phase II Cisplatin-pemetrexed Cediranib 20mg | Phase II Cisplatin-pemetrexed Placebo
All-Cause Mortality (participants affected / at risk) | 7/7 | 9/13 | 39/45 | 41/47
Serious Adverse Events (participants affected / at risk) | 4/7 | 6/13 | 32/44 | 25/46
Other Adverse Events (participants affected / at risk) | 7/7 | 13/13 | 42/44 | 43/46
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase I Cisplatin-pemetrexed Cediranib 30mg (N=7) | Phase I Cisplatin-pemetrexed Cediranib 20mg (N=13) | Phase II Cisplatin-pemetrexed Cediranib 20mg (N=44) | Phase II Cisplatin-pemetrexed Placebo (N=46)
Anemia (Blood and lymphatic system disorders) | 0 | 1 | 1 | 5
Acute coronary syndrome (Cardiac disorders) | 0 | 0 | 0 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 1 | 2 | 1
Atrial flutter (Cardiac disorders) | 0 | 0 | 1 | 1
Heart failure (Cardiac disorders) | 0 | 1 | 2 | 1
Mobitz (type) II atrioventricular block (Cardiac disorders) | 0 | 0 | 1 | 0
Pericardial effusion (Cardiac disorders) | 0 | 0 | 1 | 1
Pericarditis (Cardiac disorders) | 0 | 0 | 0 | 1
Sinus bradycardia (Cardiac disorders) | 0 | 0 | 2 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 1 | 0
Supraventricular tachycardia (Cardiac disorders) | 0 | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Ascites (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Diarrhea (Gastrointestinal disorders) | 1 | 1 | 0 | 0
Duodenal hemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Gastrointestinal disorders-Other (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Ileus (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 2 | 1 | 2
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Vomiting (Gastrointestinal disorders) | 0 | 2 | 0 | 1
Fatigue (General disorders) | 0 | 0 | 1 | 0
General disorders and admin site conditions - Other (General disorders) | 0 | 0 | 0 | 1
Localized edema (General disorders) | 1 | 0 | 0 | 0
Malaise (General disorders) | 0 | 0 | 0 | 1
Non-cardiac chest pain (General disorders) | 0 | 0 | 2 | 0
Pain (General disorders) | 0 | 1 | 0 | 0
Sudden death NOS (General disorders) | 0 | 0 | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 1 | 0
Appendicitis perforated (Infections and infestations) | 0 | 0 | 1 | 0
Lung infection (Infections and infestations) | 0 | 2 | 1 | 4
Sepsis (Infections and infestations) | 0 | 0 | 1 | 0
Soft tissue infection (Infections and infestations) | 0 | 0 | 1 | 0
Upper respiratory infection (Infections and infestations) | 0 | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Wound dehiscence (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Blood bilirubin increased (Investigations) | 1 | 0 | 0 | 0
Cardiac troponin I increased (Investigations) | 0 | 0 | 1 | 0
Creatinine increased (Investigations) | 0 | 0 | 1 | 0
Lymphocyte count decreased (Investigations) | 0 | 0 | 1 | 0
Neutrophil count decreased (Investigations) | 0 | 0 | 2 | 2
Platelet count decreased (Investigations) | 0 | 0 | 2 | 0
Weight loss (Investigations) | 0 | 0 | 1 | 0
White blood cell decreased (Investigations) | 0 | 0 | 2 | 2
Anorexia (Metabolism and nutrition disorders) | 0 | 0 | 3 | 2
Dehydration (Metabolism and nutrition disorders) | 0 | 3 | 5 | 1
Hypocalcemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Hypokalemia (Metabolism and nutrition disorders) | 0 | 0 | 2 | 0
Hypomagnesemia (Metabolism and nutrition disorders) | 0 | 0 | 2 | 0
Hyponatremia (Metabolism and nutrition disorders) | 0 | 0 | 5 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1
Neoplasms benign, malignant and unspecified - Other (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 3 | 4
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 1
Intracranial hemorrhage (Nervous system disorders) | 0 | 0 | 1 | 0
Nervous system disorders-Other (Nervous system disorders) | 0 | 1 | 0 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 0 | 0 | 1
Seizure (Nervous system disorders) | 0 | 0 | 1 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 1
Transient ischemic attacks (Nervous system disorders) | 0 | 0 | 1 | 0
Confusion (Psychiatric disorders) | 0 | 1 | 2 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 1 | 0
Chronic kidney disease (Renal and urinary disorders) | 0 | 0 | 1 | 0
Renal and urinary disorders-Other (Renal and urinary disorders) | 0 | 0 | 0 | 1
Urinary retention (Renal and urinary disorders) | 0 | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1 | 3
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 3 | 0
Hypertension (Vascular disorders) | 0 | 0 | 1 | 0
Hypotension (Vascular disorders) | 0 | 0 | 3 | 0
Thromboembolic event (Vascular disorders) | 0 | 0 | 5 | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Phase I Cisplatin-pemetrexed Cediranib 30mg (N=7) | Phase I Cisplatin-pemetrexed Cediranib 20mg (N=13) | Phase II Cisplatin-pemetrexed Cediranib 20mg (N=44) | Phase II Cisplatin-pemetrexed Placebo (N=46)
Anemia (Blood and lymphatic system disorders) | 7 | 10 | 30 | 31
Blood and lymphatic system disorders - Other (Blood and lymphatic system disorders) | 1 | 0 | 1 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 2 | 1 | 2
Atrial flutter (Cardiac disorders) | 1 | 0 | 0 | 1
Cardiac disorders-Other (Cardiac disorders) | 0 | 1 | 1 | 0
Chest pain - cardiac (Cardiac disorders) | 1 | 1 | 0 | 0
Mitral valve disease (Cardiac disorders) | 1 | 0 | 0 | 0
Palpitations (Cardiac disorders) | 1 | 0 | 1 | 0
Pericardial effusion (Cardiac disorders) | 2 | 0 | 0 | 1
Pericarditis (Cardiac disorders) | 1 | 0 | 0 | 0
Restrictive cardiomyopathy (Cardiac disorders) | 1 | 0 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 1 | 0 | 2 | 1
Ear pain (Ear and labyrinth disorders) | 1 | 0 | 0 | 0
Hearing impaired (Ear and labyrinth disorders) | 0 | 2 | 4 | 6
Tinnitus (Ear and labyrinth disorders) | 0 | 2 | 6 | 3
Endocrine disorders-Other (Endocrine disorders) | 3 | 2 | 2 | 0
Hypothyroidism (Endocrine disorders) | 2 | 2 | 10 | 3
Blurred vision (Eye disorders) | 0 | 0 | 3 | 0
Dry eye (Eye disorders) | 1 | 0 | 0 | 1
Watering eyes (Eye disorders) | 0 | 0 | 1 | 5
Abdominal distension (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 3 | 5 | 2 | 5
Bloating (Gastrointestinal disorders) | 0 | 2 | 0 | 0
Cheilitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 7 | 8 | 21 | 21
Diarrhea (Gastrointestinal disorders) | 5 | 8 | 22 | 9
Dry mouth (Gastrointestinal disorders) | 1 | 0 | 4 | 2
Dyspepsia (Gastrointestinal disorders) | 1 | 1 | 7 | 3
Dysphagia (Gastrointestinal disorders) | 0 | 2 | 3 | 2
Esophageal pain (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Gastritis (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 | 3 | 5 | 0
Gastrointestinal disorders-Other (Gastrointestinal disorders) | 1 | 4 | 2 | 0
Gastroparesis (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Mucositis oral (Gastrointestinal disorders) | 3 | 2 | 7 | 8
Nausea (Gastrointestinal disorders) | 6 | 12 | 32 | 30
Oral pain (Gastrointestinal disorders) | 1 | 1 | 3 | 0
Rectal hemorrhage (Gastrointestinal disorders) | 1 | 0 | 2 | 0
Toothache (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 5 | 11 | 14 | 14
Chills (General disorders) | 0 | 1 | 1 | 0
Edema limbs (General disorders) | 3 | 2 | 5 | 6
Edema trunk (General disorders) | 1 | 0 | 0 | 1
Fatigue (General disorders) | 7 | 12 | 33 | 34
Fever (General disorders) | 0 | 0 | 4 | 3
General disorders and admin site conditions - Other (General disorders) | 0 | 1 | 0 | 2
Non-cardiac chest pain (General disorders) | 1 | 5 | 16 | 9
Pain (General disorders) | 3 | 5 | 6 | 2
Cholecystitis (Hepatobiliary disorders) | 1 | 0 | 0 | 1
Gallbladder obstruction (Hepatobiliary disorders) | 1 | 0 | 1 | 0
Allergic reaction (Immune system disorders) | 1 | 2 | 0 | 0
Infections and infestations-Other (Infections and infestations) | 0 | 2 | 0 | 0
Mucosal infection (Infections and infestations) | 0 | 0 | 0 | 3
Pleural infection (Infections and infestations) | 1 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 2 | 0 | 1 | 1
Soft tissue infection (Infections and infestations) | 1 | 0 | 0 | 0
Tooth infection (Infections and infestations) | 1 | 1 | 0 | 1
Upper respiratory infection (Infections and infestations) | 1 | 1 | 2 | 2
Urinary tract infection (Infections and infestations) | 4 | 2 | 6 | 5
Bruising (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 2
Activated partial thromboplastin time prolonged (Investigations) | 1 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 4 | 1 | 5 | 4
Alkaline phosphatase increased (Investigations) | 3 | 2 | 6 | 7
Aspartate aminotransferase increased (Investigations) | 5 | 2 | 9 | 6
Blood bilirubin increased (Investigations) | 2 | 3 | 1 | 3
Cholesterol high (Investigations) | 3 | 3 | 5 | 2
Creatinine increased (Investigations) | 1 | 6 | 12 | 15
INR increased (Investigations) | 1 | 0 | 1 | 0
Investigations-Other (Investigations) | 1 | 1 | 1 | 2
Lymphocyte count decreased (Investigations) | 5 | 0 | 8 | 10
Neutrophil count decreased (Investigations) | 5 | 8 | 18 | 17
Platelet count decreased (Investigations) | 3 | 6 | 13 | 10
Weight loss (Investigations) | 4 | 8 | 19 | 13
White blood cell decreased (Investigations) | 6 | 5 | 18 | 14
Anorexia (Metabolism and nutrition disorders) | 6 | 8 | 23 | 17
Dehydration (Metabolism and nutrition disorders) | 2 | 3 | 10 | 13
Glucose intolerance (Metabolism and nutrition disorders) | 3 | 2 | 3 | 1
Hypercalcemia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 1
Hyperglycemia (Metabolism and nutrition disorders) | 0 | 3 | 16 | 13
Hyperkalemia (Metabolism and nutrition disorders) | 0 | 5 | 7 | 14
Hypernatremia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Hypertriglyceridemia (Metabolism and nutrition disorders) | 0 | 1 | 1 | 1
Hyperuricemia (Metabolism and nutrition disorders) | 0 | 2 | 2 | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 6 | 4 | 15 | 15
Hypocalcemia (Metabolism and nutrition disorders) | 2 | 4 | 10 | 6
Hypoglycemia (Metabolism and nutrition disorders) | 0 | 2 | 2 | 3
Hypokalemia (Metabolism and nutrition disorders) | 1 | 5 | 7 | 10
Hypomagnesemia (Metabolism and nutrition disorders) | 6 | 9 | 21 | 17
Hyponatremia (Metabolism and nutrition disorders) | 4 | 5 | 20 | 18
Hypophosphatemia (Metabolism and nutrition disorders) | 0 | 2 | 2 | 1
Metabolism and nutrition disorders - Other, specify (Metabolism and nutrition disorders) | 2 | 4 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 0 | 1 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 5 | 4 | 3
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 4 | 1
Chest wall pain (Musculoskeletal and connective tissue disorders) | 3 | 5 | 6 | 6
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 | 4 | 9 | 5
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Musculoskeletal and connective tiss disorder - Other (Musculoskeletal and connective tissue disorders) | 3 | 0 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 1 | 3 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 1 | 6 | 2
Ataxia (Nervous system disorders) | 0 | 2 | 0 | 0
Cognitive disturbance (Nervous system disorders) | 1 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 2 | 3 | 5 | 6
Dysgeusia (Nervous system disorders) | 2 | 1 | 12 | 5
Headache (Nervous system disorders) | 2 | 3 | 7 | 3
Memory impairment (Nervous system disorders) | 0 | 1 | 1 | 0
Paresthesia (Nervous system disorders) | 0 | 1 | 2 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 1 | 3 | 11 | 9
Presyncope (Nervous system disorders) | 0 | 1 | 1 | 0
Tremor (Nervous system disorders) | 0 | 0 | 3 | 0
Anxiety (Psychiatric disorders) | 2 | 5 | 7 | 7
Confusion (Psychiatric disorders) | 0 | 1 | 1 | 2
Depression (Psychiatric disorders) | 0 | 4 | 7 | 3
Insomnia (Psychiatric disorders) | 5 | 2 | 7 | 5
Psychiatric disorders-Other (Psychiatric disorders) | 1 | 0 | 2 | 0
Hematuria (Renal and urinary disorders) | 1 | 0 | 3 | 0
Proteinuria (Renal and urinary disorders) | 6 | 10 | 17 | 5
Renal and urinary disorders-Other (Renal and urinary disorders) | 2 | 0 | 1 | 0
Urinary frequency (Renal and urinary disorders) | 0 | 2 | 0 | 3
Urinary incontinence (Renal and urinary disorders) | 0 | 1 | 1 | 0
Urinary retention (Renal and urinary disorders) | 1 | 0 | 1 | 1
Irregular menstruation (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Prostatic obstruction (Reproductive system and breast disorders) | 3 | 0 | 4 | 0
Prostatic pain (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 5 | 0
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 6 | 15 | 9
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 4 | 11 | 23 | 16
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 7 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 4
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 4 | 3 | 3 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 4 | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 1 | 0
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 2 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 3 | 4
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Resp, thoracic and mediastinal disorders - Other (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
Sleep apnea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
Sore throat (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2 | 2
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 6 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 1 | 2 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 1 | 3 | 2
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 2 | 2 | 1
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 1 | 0 | 2 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1 | 2 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 3 | 4 | 4
Skin and subcutaneous tissue disorders - Other (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 2
Hot flashes (Vascular disorders) | 0 | 1 | 0 | 0
Hypertension (Vascular disorders) | 4 | 9 | 25 | 12
Hypotension (Vascular disorders) | 1 | 0 | 2 | 5
Thromboembolic event (Vascular disorders) | 0 | 1 | 1 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-01-05): https://cdn.clinicaltrials.gov/large-docs/48/NCT01064648/Prot_SAP_000.pdf